CLINICAL TRIAL: NCT05066646
Title: Phase 1/2 Clinical Study on Fully Human BCMA Chimeric Antigen Receptor Autologous T Cell Injection (CT103A) in the Treatment of Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Phase 1/2 Study of a Fully Human BCMA-targeting CAR (CT103A) in Patients With Relapsed/Refractory Multiple Myeloma (FUMANBA-1)
Acronym: FUMANBA-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL-LCYJ-0007
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — CT103A chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT103A in relapsed and refractory multiple myeloma patients (Experimental): CT103A autologous CAR-T cells will be infused at RP2D of 1.0 x 10^6 CAR+ T cells after receiving lymphodepleting chemotherapy
  Interventions: Drug: CT103A

INTERVENTIONS:
Drug: CT103A — CT103A consists of autologous T lymphocytes transduced with anti-BCMA CAR lentiviral vector that containing a unique CAR structure with a fully human single-chain variable fragment (scFv).

SUMMARY:
This study is a single-armed, open-label, multicenter Phase 1/2 study to evaluate the efficacy and safety of CT103A in subjects with relapsed and refractory MM.

DETAILED DESCRIPTION:
Leukapheresis procedure will be performed to manufacture CT103A chimeric antigen receptor (CAR) modified T cells. Bridging therapy is allowed between PBMC collection and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. After 1-day rest, subjects will receive a single dose infusion of CT103A at 1.0 x 10^6 CAR+ T cells/Kg. Subjects will be followed in the study for a minimum of 2 years after CT103A infusion. Long-term follow-up for lentiviral vector safety will be followed for up to 15 years after CT103A infusion.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all the following criteria to be enrolled in the study:

1. age 18 to 70 years old, male or female.
2. Subjects with diagnosed relapsed or refractory MM according to IMWG criteria and have had at least 3 prior lines of therapy including chemotherapy based on proteasome inhibitors (PIs) and immunomodulatory agents (IMiDs). Disease progression must be documented during or within 12 months following the most recent anti-myeloma treatment.
3. Evidence of cell membrane BCMA expression, as determined by a validated immunohistochemistry (IHC) or flow cytometry of tumor tissue (e.g., bone marrow biopsies, or plasmacytoma).
4. The subjects should have measurable disease based on at least one of the following parameters:

   * The proportion of primitive immature or monoclonal plasma cells detected by bone marrow cytology, bone marrow biopsy, or flow cytometry is ≥ 5%.
   * Serum M-protein ≥ 0.5 g/dL.
   * Urine M-protein ≥ 200 mg/24 hrs.
   * For those whose Serum or Urine M-protein does not meet the measurable criteria but the light chain type, serum free light chain (sFLC): involved sFLC level ≥ 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal.
5. ECOG performance score 0-1.
6. Estimated life expectancy ≥ 12 weeks.
7. Patients should have adequate organ function:

   * Hematology: Absolute neutrophil count (ANC) ≥1×10^9 /L (prior use of growth factor support is permitted, but subjects must not have received supportive treatment within 7 days prior to laboratory examination); absolute lymphocyte count (ALC) ≥0.3×10^9 /L; platelets ≥50×10^9 /L (subjects must not have received blood transfusion support within 7 days prior to laboratory examination); hemoglobin ≥60 g/L (subjects must not have received transfusion of red blood cells [RBC] within 7 days prior to laboratory examination; the use of recombinant human erythropoietin is permitted).
   * Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×upper limit of normal (ULN); total serum bilirubin ≤ 1.5×ULN.
   * Renal function: Creatinine clearance rate (CrCl) calculated according to Cockcroft-Gault formula ≥ 40 ml/min.
   * Coagulation function: Fibrinogen ≥ 1.0 g/L; activated partial thromboplastin time (APTT) ≤ 1.5×ULN, prothrombin time (PT) ≤ 1.5×ULN.
   * SpO2 > 91%.
   * Left ventricular ejection fraction (LVEF) ≥ 50%.
8. The subject and his/her spouse agree to use an effective contraceptive tool or medication (excluding safety period contraception) for one year from the date of the subject's informed consent to the date of CAR T cell infusion.
9. Subject must sign the informed consent form approved by ethics board in person before starting any screening procedure.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subjects who are known to have GVHD or need long-term immunosuppressive therapy.
2. Subjects have received an autologous hematopoietic stem cell transplantation (auto-HSCT) within 12 weeks before leukapheresis or have a previous history of two times of allo-HSCT or previous history of an allogeneic hematopoietic stem cell transplantation (allo-HSCT).
3. Insufficient mononuclear cells for CAR T cell production.
4. Subjects have received any anti-cancer treatment as follows: targeted therapies, epigenetic therapy or invasive experimental instruments therapy within 14 days or at least 5 half-lives before leukapheresis (according to the longer time), or monoclonal antibody for treating multiple myeloma within 21 days before leukapheresis, or cytotoxic therapy or proteasome inhibitors within 14 days before leukapheresis, or immunomodulatory agents within 7 days before leukapheresis.
5. Subjects who were receiving a used therapeutic dose of corticosteroid treatment (defined as prednisone or equivalent > 20mg) within 7 days prior to screening, except for physiological alternatives, inhalation, or topical use.
6. Subjects with serious heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmias.
7. Subjects with systemic diseases that the investigator determined to be unstable include, but are not limited to, severe liver and kidney or metabolic diseases requiring medical treatment.
8. Subjects with second malignancies in addition to MM within the past 5 years before the screening, exceptions to this criterion: successfully treated cervical carcinoma in situ and non-metastatic basal or squamous cell skin carcinoma, local prostate cancer after radical surgery, and ductal carcinoma in situ of the breast after radical surgery.
9. Subjects with a history of organ transplantation.
10. Subjects have central nervous system (CNS) involvement (including cranial neuropathies or mass lesions and leptomeningeal disease).
11. Subjects with extramedullary lesions (except for a single extramedullary lesion with a maximum transverse diameter of 3 cm).
12. Subjects with plasma cell leukemia.
13. Subjects have received major surgery within 2 weeks prior to leukapheresis or plan to receive surgery during the study or within 2 weeks after the study treatment (excluding local anesthesia).
14. Subjects participated in another interventional clinical study 3 months before signing the informed consent (ICF);
15. Subjects with any uncontrolled active infection needed to receive systemic therapy within 7 days before leukapheresis collection (excluding < CTCAE grade 2 urogenital infection and upper respiratory infection).
16. Positive for any of the following tests:

    * Hepatitis B virus (HBV) surface antigen (HBsAg) or hepatitis B core antibody-positive and detectable HBV DNA in peripheral blood
    * Hepatitis C virus (HCV) antibody and hepatitis C virus RNA in peripheral blood
    * Human immunodeficiency virus (HIV) antibody
    * Cytomegalovirus (CMV) DNA
    * Treponema Pallidum antibody
17. Pregnant or lactating women.
18. Subjects with mental illness or consciousness disorder or disease of the central nervous system
19. Subjects who haven't recovery to Grade 1 or baseline of any toxicities due to prior treatments, excluding alopecia.
20. Other conditions that researchers consider inappropriate for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence and Severity of Adverse Events | Minimum of 2 years post CT103A infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Phase 1: Laboratoty tests | Minimum of 2 years post CT103A infusion
  Abnormal results of laboratoty tests
Phase 1: Vital signs | Minimum of 2 years post CT103A infusion
  Abnormal results of vital signs
Phase 1: Physical examination | Minimum of 2 years post CT103A infusion
  Abnormal results of physical examination
Phase 2: Overall response rate (ORR) evaluated by an Independent Review Committee (IRC) | 3 months post CT103A infusion
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by an IRC

SECONDARY OUTCOMES:
Overall response rate (ORR) evaluated by the investigators | 3 months post CT103A infusion
  Percentage of subjects who achieved partial response (PR) or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by the investigators
Overall Survival (OS) | Minimum of 2 years post CT103A infusion
  Time from CT103A infusion to time of death due to any cause
Duration of Response (DOR) | Minimum of 2 years post CT103A infusion
  Time from first response evaluated by an IRC or investigators to disease progression or death from any cause
Progression-free Survival (PFS) | Minimum of 2 years post CT103A infusion
  Time from CT103A infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first
Time to Response (TTR) | Minimum of 2 years post CT103A infusion
  Time from CT103A infusion to first documentation of response evaluated by an IRC or investigators
Laboratoty tests | Minimum of 2 years post CT103A infusion
  Abnormal results of laboratoty tests
Vital signs | Minimum of 2 years post CT103A infusion
  Abnormal results of vital signs
Physical examination | Minimum of 2 years post CT103A infusion
  Abnormal results of physical examination
Minimal Residual Disease (MRD) | Minimum of 2 years post CT103A infusion
  Proportion of subjects who achieved MRD negative
Pharmacokinetics - Cmax | Minimum of 2 years post CT103A infusion
  The maximum transgene level at Tmax
Pharmacokinetics - Tmax | Minimum of 2 years post CT103A infusion
  Time to peak transgene level
Pharmacokinetics - AUC0-28days | Minimum of 2 years post CT103A infusion
  Area under the curve of CAR T cells from time zero to Day 28
Pharmacokinetics - AUC0-90days | Minimum of 2 years post CT103A infusion
  Area under the curve of CAR T cells from time zero to Day 90
soluble BCMA levels | Minimum of 2 years post CT103A infusion
  soluble BCMA levels in peripheral blood of subjects

OTHER OUTCOMES:
Immunogenicity | Minimum of 2 years post CT103A infusion
  Development of an anti-CAR antibody response
replication competent lentivirus (RCL) | Minimum of 2 years post CT103A infusion
  The incidence of replication competent lentivirus (RCL)
the levels of CAR-T related inflammatory factors | Minimum of 2 years post CT103A infusion
  the levels of CRP, IL-6 and Ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MD, PhD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Chunrui Li, MD, PhD, Principal Investigator — Tongji Hospital
Locations (14):
- China (14):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The Affiliated Cancer Hospital of Zhengzhou University and Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Boren Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Xinqiao Hospital, Army Medical University, Chongqing
  - Fudan University Zhongshan Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keam SJ. Equecabtagene Autoleucel: First Approval. Mol Diagn Ther. 2023 Nov;27(6):781-787. doi: 10.1007/s40291-023-00673-y. Epub 2023 Sep 2. PMID 37658205
- [Derived] Zhou L, Fu W, Wu S, Xu K, Qiu L, Xu Y, Yan X, Zhang Q, Zhang M, Wang L, Hong R, Chang AH, Yu J, Fu S, Kong D, Li L, Wang Y, Li Z, Jiang H, Huang J, Liu Z, Su N, Wei G, Hu Y, Huang H. Derivation and validation of a novel score for early prediction of severe CRS after CAR-T therapy in haematological malignancy patients: A multi-centre study. Br J Haematol. 2023 Aug;202(3):517-524. doi: 10.1111/bjh.18873. Epub 2023 May 16. PMID 37192741